CLINICAL TRIAL: NCT07365605
Title: INTERACTION BETWEEN MUSCLE MASS AND BALANCE PERFORMANCE: A LOWER-LIMB-FOCUSED ANALYSIS
Brief Title: Lower-Limb Muscle Mass and Balance Performance
Acronym: LMBP
Status: Not yet recruiting | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Ramiz ARABACI, Principal Investigator, Uludag University
Other Study IDs: E-87914409-050.04-117156
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Lower-limb Muscle Mass and Balance Performance
Keywords: Balance performance; Relative muscle mass; Lower-limb muscles; Postural stability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower Balance Performance Group (LBP): This cohort will include moderately physically active young men who exhibit higher sway path length values during a 30-second center-of-pressure-based static balance test, indicating lower balance performance. Participants in this group will have no musculoskeletal, neurological, or medical conditions affecting postural control. This cohort will be used to examine muscle mass characteristics associated with relatively poorer balance performance.
- Higher Balance Performance Group (HBP): This cohort will include moderately physically active young men who exhibit lower sway path length values during a 30-second center-of-pressure-based static balance test, indicating higher balance performance. Participants in this group will be free from conditions that may influence balance outcomes. This cohort will be used to evaluate muscle mass characteristics associated with relatively better balance performance.

SUMMARY:
This study will examine the interaction between lower-limb muscle mass and balance performance in moderately physically active young men. Body composition parameters, including appendicular skeletal muscle mass, leg muscle mass, and the ratio of lower-limb muscle mass to body weight (LMM/BW), will be assessed using bioelectrical impedance analysis. Balance performance will be evaluated using a center-of-pressure-based static balance test, with classifications derived from sway path length and sway area parameters.

Participants will be grouped according to balance performance metrics, and muscle mass indicators will be compared between balance-based groups. Correlation analyses will also be conducted to explore associations between muscle mass variables and balance outcomes across the entire sample. It is anticipated that normalized muscle mass indicators, particularly LMM/BW, will demonstrate greater discriminative sensitivity than absolute muscle mass measures in relation to balance performance. The findings are expected to contribute to a more precise understanding of how relative lower-limb muscular capacity relates to postural control in young, physically active populations.

DETAILED DESCRIPTION:
This study will employ a cross-sectional observational design to investigate the relationship between lower-limb muscle mass and balance performance in moderately physically active young men. The primary focus will be to determine whether normalized muscle mass indicators, particularly the ratio of lower-limb muscle mass to body weight (LMM/BW), demonstrate greater sensitivity in explaining balance-performance differences than absolute muscle mass measures.

A cohort of healthy male participants aged 20-30 years will be recruited. All participants will be moderately physically active and free from musculoskeletal injuries, neurological disorders, or medical conditions that could affect balance performance. After providing written informed consent, participants will undergo standardized anthropometric and body composition assessments using bioelectrical impedance analysis to obtain appendicular skeletal muscle mass, leg muscle mass, total muscle mass, body fat percentage, and LMM/BW.

Balance performance will be evaluated using a center-of-pressure-based static balance test performed on a stabilometric platform. Participants will complete a 30-second quiet standing task, during which sway path length and sway area will be recorded as primary balance outcomes. These parameters will be used to classify participants into balance-performance-based groups in order to examine the discriminative capacity of different balance metrics with respect to muscle mass variables.

Between-group comparisons of muscle mass indicators will be conducted to identify differences associated with balance performance classifications. In addition, correlation analyses will be performed across the entire sample to assess the strength and direction of associations between muscle mass variables and balance outcomes. Effect size estimates will be calculated to support the interpretation of observed differences.

The study is expected to clarify whether relative lower-limb muscular capacity provides a more functionally meaningful explanation of balance performance than absolute muscle mass in young, physically active populations. The findings may contribute to improved methodological approaches in balance assessment and support the use of normalized muscle mass indicators in sports science, exercise physiology, and preventive health contexts.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria required that participants (i) were between 20 and 30 years of age; (ii) had no lower-limb injuries that could affect test performance; (iii) were moderately physically active; and (iv) had not used ergogenic aids or stimulant substances for at least six months prior to the study.

Exclusion Criteria:

* Exclusion criteria included the presence of back, neck, leg, foot, or upper-limb pain within the previous six months, as well as a history of major orthopedic surgery involving the lower extremities or trunk.

Ages: 20 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eskisehir, TURKEY
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Balance performance assessed by center-of-pressure sway path length | Day 1 (Assessed during a single laboratory testing session)
  Balance performance will be quantified using center-of-pressure sway path length recorded during a 30-second quiet standing test on a stabilometric platform. Sway path length will represent the total displacement of the center of pressure over the trial duration, with higher values indicating poorer balance performance. This measure will serve as the primary balance outcome for group classification and for association analyses with lower-limb muscle mass indicators.

IPD SHARING:
Plan to Share IPD: No
This study will use a cross-sectional observational design to examine the relationship between lower-limb muscle mass and balance performance in moderately physically active young men. Participants will complete standardized body composition assessments and a center-of-pressure-based static balance test during a single laboratory visit. Based on sway path length values, participants will be classified into lower and higher balance performance groups.
  Comparisons of muscle mass indicators, including absolute and normalized measures, will be conducted between balance-performance-based groups. In addition, associations between muscle mass variables and balance outcomes will be analyzed across the full sample to evaluate the relative explanatory value of different muscle mass indicators. The study plan is intended to determine whether normalized lower-limb muscle mass measures provide greater sensitivity for explaining balance performance differences than absolute muscle mass measures.

REFERENCES:
- [Background] Lesinski M, Hortobagyi T, Muehlbauer T, Gollhofer A, Granacher U. Effects of Balance Training on Balance Performance in Healthy Older Adults: A Systematic Review and Meta-analysis. Sports Med. 2015 Dec;45(12):1721-38. doi: 10.1007/s40279-015-0375-y. PMID 26325622
- [Background] Granacher, U., Gollhofer, A., & Hortobágyi, T. (2013). Effects of strength training on balance ability in older adults: A systematic review and meta-analysis. Sports Medicine, 43(6), 515-529. https://doi.org/10.1007/s40279-013-0045-y
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Calbet JA, Radegran G, Boushel R, Saltin B. On the mechanisms that limit oxygen uptake during exercise in acute and chronic hypoxia: role of muscle mass. J Physiol. 2009 Jan 15;587(2):477-90. doi: 10.1113/jphysiol.2008.162271. Epub 2008 Dec 1. PMID 19047206
- [Background] Bohannon RW, Bubela DJ, Magasi SR, Wang YC, Gershon RC. Sit-to-stand test: Performance and determinants across the age-span. Isokinet Exerc Sci. 2010;18(4):235-240. doi: 10.3233/IES-2010-0389. PMID 25598584